CLINICAL TRIAL: NCT04746326
Title: Operative and Conservative Treatment in Right Colon Diverticulitis Patients
Brief Title: Treatment in Right Colon Diverticulitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Semra Demirli Atici, Primary investigator, Tepecik Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020 / 14-6
Record Dates: First submitted 2021-01-29; First posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Outcome
Keywords: diverticulum; surgery; appendicitis; sigmoid volvulus; caecum; diverticulitis
MeSH Terms: conditions — Diverticulum; Appendicitis; Diverticulitis | interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Conservative treatment, Operative treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conservative treatment (Other): Conservative treatment stopping oral intake, intravenous antibiotic therapy.
  Interventions: Other: Conservative treatment
- Operative treatment (Other): Operative procedure Right hemicolectomy Wedge resection of cecum Diverticulectomy + appendectomy Diverticulectomy Appendectomy + drainage
  Interventions: Procedure: Failure conservative treatment; Procedure: Surgery

INTERVENTIONS:
Procedure: Failure conservative treatment — Surgery was performed in patients who failed conservative treatment.
  Arms: Operative treatment
Procedure: Surgery — Surgery was performed in patients who had generalized peritonitis and perforation.
  Arms: Operative treatment
Other: Conservative treatment — Conservative treatment was performed in patients who had no generalized peritonitis and perforation.
  Arms: Conservative treatment

SUMMARY:
The right colon diverticula, unlike those in the left colon, contain all layers of the colon and is called the true diverticulum. Perforation is observed less frequently due to its full thickness. Conservative treatment can be applied unless complications such as abscess formation and free perforation occur. Unlike the left, right colon diverticulitis has low complications and can be treated conservatively. The differential diagnosis of right colon diverticulitis should be kept in mind in order to prevent unnecessary surgeries. Surgical treatment is inevitable in cases such as recurrent diverticulitis, generalized peritonitis, and suspected malignancy.

DETAILED DESCRIPTION:
The right colon diverticula, unlike those in the left colon, contain all layers of the colon and is called the true diverticulum. Perforation is observed less frequently due to its full thickness. Conservative treatment can be applied unless complications such as abscess formation and free perforation occur. Here, we aimed to discuss the results of conservative and surgical treatment for right colon diverticulitis in the light of the literature. 150 patients treated for colon diverticulitis between 2015-2020 were retrospectively screened. Right colon diverticulitis detected incidentally, missing data, and left colon diverticulitis were excluded from the study. Data of a total of 26 patients were accessed. Unlike the left, right colon diverticulitis has low complications and can be treated conservatively. The differential diagnosis of right colon diverticulitis should be kept in mind in order to prevent unnecessary surgeries. Surgical treatment is inevitable in cases such as recurrent diverticulitis, generalized peritonitis, and suspected malignancy

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with right colon diverticulitis

Exclusion Criteria:

* Left colon diverticulitis
* Right colon diverticulitis detected incidentally
* lacking data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with mortality | up to 24 weeks
  mortality
Number of Participants with wound infection | up to 24 weeks
  wound infection

CONTACTS AND LOCATIONS:
Locations (1):
- Tepecik Training and Research Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No